CLINICAL TRIAL: NCT05695469
Title: The Impact of Smart Resuscitation Glove (ResuGlove) as Chest Compression Feedback Devices During CPR Training: Feasibility Study of the Device Under Development
Brief Title: The Impact of ResuGlove as a Chest Compression Feedback Device
Acronym: ResuGlove
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Aalto University (Other)
Responsible Party: Principal Investigator, Desale Tewelde Kahsay, Doctoral researcher, University of Turku
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TY/739/2022
Record Dates: First submitted 2022-12-01; First posted 2023-01-25 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Testing, Reality
Keywords: Smart glove; CPR training; Sensibility study; Realtime feedback

STUDY DESIGN:
Intervention Model Description: The randomly selected participants will be randomly assigned into two equal groups using the online-based random number generator (https://www.random.org). In the first round, group 1 will perform hand-only CPR wearing the ResuGlove with a running feedback program for 2 minutes. On the other hand, group 2 will perform the same way as group 1, but without ResuGlove. After 30 minutes of recovery, in the second round, they will crossover. Ultimately, we will ask participants to fill out the SUS questionnaire.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ResuGlove group (Experimental): Participants in the ResuGlove group will be guided by the audio feedback from the smart resuscitation glove.
  Interventions: Device: Smart resuscitation glove (ResuGlove); Other: Traditional CPR
- Traditional CPR group (Active Comparator): Participants in the traditional CPR group will perform chest compressions without guidance from the smart resuscitation glove.
  Interventions: Device: Smart resuscitation glove (ResuGlove); Other: Traditional CPR

INTERVENTIONS:
Device: Smart resuscitation glove (ResuGlove) — Participants will be randomly assigned into two equal groups using the online-based random number generator (https://www.random.org). Participants in the ResuGlove group will perform hand-only CPR wearing the ResuGlove with a running feedback program for 2 minutes.
Other: Traditional CPR — Participants in the traditional CPR group will perform hand-only CPR without the ResuGlove and feedback guidance for 2 minutes.

SUMMARY:
The goal of this simulation-based randomized trial is to assess if the newly proposed ResuGlove can improve the quality of chest compressions during CPR training of laypersons and inexperienced health professionals. The main questions it aims to answer are:

1. To determine if the newly developed wearable resuscitation gloves will improve the quality of chest compression during simulation-based CPR training
2. To determine the learnability and usability of the ResuGlove using the System Usability Scale (SUS) questionnaire

Participants will be randomly assigned into two equal groups the ResuGlove group (group 1) vs the traditional CPR group (Group 2). The investigators will compare the quality of chest compression between these two groups. On the same day, participants will be asked about the learnability and usability of ResuGlove using the System Usability Scale (SUS questionnaire.

DETAILED DESCRIPTION:
AIM OF THE STUDY:

This study is part of an upgoing project to develop smart resuscitation gloves (ResuGlove) that help evaluate the quality of chest compressions during CPR training. The ResuGlove are smart-textile-based wearable technologies expected to provide real-time audiovisual feedback on chest compression quality, including compression depth, compression rate and chest recoil.

This feasibility study aims to evaluate if the newly proposed ResuGloves can significantly improve the quality of chest compressions compared to traditional CPR during simulated cardiac arrest. Besides, researchers will evaluate the learnability and usability of ResuGloves using the System Usability Scale (SUS) questionnaire.

HYPOTHESIS:

Hypothesis 1: ResuGlove will significantly improve the quality of chest compressions compared to the traditional CPR during simulated cardiac arrest Hypothesis 2: Research participants will positively rate the learnability and usability of the ResuGloves under development.

SIGNIFICANCE OF THE STUDY:

To begin with, the result of this preliminary feasibility study will guide the researchers on device modification and future design. Besides, this feasibility study will help researchers design a more extensive controlled trial study to compare the newly developed devices with similar feedback devices during laypersons' CPR training. Once the ResuGloves are fully developed and implemented, they will be used to train laypersons in communities. Furthermore, the currently proposed affordable and easy-to-use textile-based ResuGloves will be used to train health professionals in resource-limited settings. Finally, this study will open the door for further studies to look for other health benefits of smart gloves.

METHOD:

The investigators will use a prospective randomized controlled crossover trial of two groups to collect data on the chest compression parameters. In the first round, group 1 will perform hand-only CPR with the help of feedback from the ResuGloves, and group 2 will perform hand-only CPR without the ResuGlove. After 30 minutes of recovery, participants will crossover. Besides, participants will be asked about the learnability and usability of the ResuGlove using the system usability scale (SUS) questionnaire.

Researchers will recruit 30 volunteered nursing students from Turku University of Applied sciences .

Researchers will announce the aim of the study to the nursing students by sending an invitation letter via their university email addresses. The invitation letter will include information about the study aim, confidentiality, inclusion/ exclusion criteria, and trial design. Students will register their interest by sending an email or SMS to the emails address or telephone numbers included in the invitation letter. Finally, a simple random sampling will be used to draw the required number of participants, using a random numbers generator software (https://www.randomizer.org/). Researchers conducted a pilot study of eight participants to detect the mean difference in compression depth between the control and the ResuGlove groups. Therefore, the sample size of the actual study (30 participants) was estimated from the pilot study with an α error of 0.05 and a power of 0.8. The investigators consulted a statistician to estimate the sample size of this feasibility crossover study.

Participants will be randomly assigned into two equal groups using the online-based random number generator (https://www.random.org). In the first round, ResuGlove group will perform hand-only CPR wearing the ResuGlove with a running feedback program for 2 minutes. On the other hand, the traditional CPR group will perform the same way as the ResuGlove group, but without the ResuGlove. After 30 minutes of recovery, in the second round, participants will crossover. Ultimately, investigators will ask participants to fill out the SUS questionnaire.

Data will be presented as mean, median and percentage as necessary. Depending on the data type, the mean difference will be analyzed using either parametric or non-parametric statistics. A p-value of < 0.05 will be the significance threshold of our data analysis.

ETHICAL MATTERS:

Participants' autonomy will be assured by allowing them to voluntarily determine their participation, including the right to withdraw at any time without explaining themselves. Participants also have the right to ask questions and refuse to give information about a specific question. In addition, participants will receive an informed consent form, the questions to be asked and a detailed information sheet before enrolment. The information sheet will describe the aim, methods, implications of the research, and the nature of the participation. The investigators will collect the participants' backgrounds, such as gender, age, CPR experience and profession. However, the investigators will not ask for sensitive personal data such as name, income, social security number, color, ethnicity, address, and location. Collected personal data will be coded pseudonymously and stored in a secured computer in the Department and the University of Turku Seafile with access only to the researchers. This way, Participants' rights to privacy, confidentiality, and anonymity will be maintained. The collected data will be deleted once the project is completed. Only outcomes of the analyzed data without personal identifiers will be published in an open-access international journal. The investigators will make every effort to ensure that no participant will be recognizable in any publication.

ELIGIBILITY:
Inclusion Criteria:

* Nursing student from Turku University of Applied Sciences
* Students have a minimum of basic life support training
* Participants should be able to understand and communicate in English

Exclusion Criteria:

* Participants must not have previous experiences in actual patient resuscitation.
* Participants who are not able to understand and communicate in English
* Students with known cardiac/pulmonary diseases, back pain, and wrist problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Average Chest compression depth | At zero time point (first round) and crossover at 30 minutes (second round)
  Chest compression depth is one of the most critical components of quality CPR. The current International Liaison Committee on Resuscitation (ILCOR) guidelines recommended a chest compression depth of 5-6 cm for improved outcomes.
Average chest compression rate | At zero time point (first round) and crossover at 30 minutes (second round)
  The compression rate is another essential component of quality CPR. The current International Liaison Committee on Resuscitation (ILCOR) guidelines recommended a chest compression rate of 100 to 1200 per minute for improved outcomes.
Proportion of chest recoil | At zero time point (first round) and crossover at 30 minutes (second round)
  Complete chest release (recoil) between each compression is essential to allow the heart to accumulate blood to be pumped during compressions. Therefore, the International Liaison Committee on Resuscitation (ILCOR) guidelines recommended complete chest recoil (100%) during CPR for a better outcome.

SECONDARY OUTCOMES:
The proportion of correct compression depth | At zero time point (first round) and crossover at 30 minutes (second round)p
  The percentage of correct compression to a depth of 5-6cm within the two minutes
The proportion of correct compression rate | At zero time point (first round) and crossover at 30 minutes (second round)
  The proportion of correct compressions to a rate of 100 to 120 per minute within the two minutes
Learnability and usability of the ResuGlove under development | At the end of the second round (30 to 40 minutes)
  Participants will be asked about the learnability and usability of ResuGlove at the end of the intervention. For the learnability and usability evaluation, we will use the System Usability Scale (SUS) questionnaire, initially developed by Brooke (1996) and modified later for various technological products. The questionnaire is quick and easy to be used by the study participants. It provides a single score on a scale understood by many people. The SUS has ten statements, in which the odd numbers are positively worded, and the negative numbers are negatively worded. The final score for the SUS will range from 0 to 100. A higher score will indicate better learnability and usability.

CONTACTS AND LOCATIONS:
Overall Officials: Desale T Kahsay, MSc, Principal Investigator — University of Turku; Sanna Salanterä, Professor, Study Chair — University of Turku
Locations (1):
- University of Turku, Turku, Southwest, Finland

IPD SHARING:
Plan to Share IPD: Yes
Only outcomes of the analyzed data without personal identifiers will be publicly available after being published in an international journal.
Time Frame: When the summary data is published and made available by the Journal
Access Criteria: Access will be possible through the Journal website. The principal investigator is ready to share additional information regarding the trail following a genuine request.